CLINICAL TRIAL: NCT02865616
Title: A Phase I, Open-Label, Single-Centre Study of the Safety and Efficacy of MET-2 in Patients With Recurrent Clostridium Difficile Infection (CDI)
Brief Title: MET-2 Clinical Study for Recurrent Clostridium Difficile Infection (CDI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NuBiyota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MET-2-101
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Clostridium Difficile Infection
Keywords: CDI; recurrent infection; MET-2; C. difficile
MeSH Terms: conditions — Clostridium Infections; Reinfection | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MET-2 Capsules (Experimental): Patients will be on vancomycin to control symptoms up until the time of the treatment.
  Initial Loading Dose: Patients will be given an initial daily loading dose of 5 g MET-2 over 2 days followed by a maintenance dose of 1.5 g over 8 days. Patients who do not experience treatment failure between Day 14 and Day 40 will be monitored until Day 130.
  Second Loading Dose: Patients experiencing treatment failure after the first dose may be offered a second, higher loading dose 10 g of MET-2 in the form of 20 MET-2 capsules per day for two days, there will not be additional daily dosing beyond the first 10 days.
  Colonoscopy: Patients failing the second loading dose of MET-2 may be offered 15 g of MET-2, equivalent to a 30 MET-2 capsule loading dose by weight, via colonoscopy..
  All patients will be followed up for 120 days after the last treatment has been received.
  Interventions: Drug: MET-2; Drug: Vancomycin

INTERVENTIONS:
Drug: MET-2 — Microbial Ecosystem Therapeutics (MET) is a new treatment approach for debilitating recurrent Clostridium difficile infection that has been developed as an alternative to fecal transplantation.
Drug: Vancomycin — Patients will be on vancomycin to control symptoms up until the time of the treatment. Patient must hold their p.o. vancomycin for 24 hours prior to receiving the first dose.

SUMMARY:
MET-2 clinical study is an Open label, single center, multiple dose pilot study of 19 patients. The study is designed to measure the resolution of diarrhea as well as the feasibility of administration and safety of MET-2 for the treatment of recurrent CDI in patients who have experienced at least two prior episodes of CDI and have developed recurrence after having completed standard-of care oral antibiotic therapy to treat CDI.

DETAILED DESCRIPTION:
Microbial Ecosystem Therapeutics (MET) is a new treatment approach for debilitating recurrent Clostridium difficile infection that has been developed as an alternative to fecal transplantation. This treatment is not a drug or biologic, but is comprised of live microbes that normally reside in the human gut of a healthy individual.The product is a defined microbial community derived from healthy donor stool, referred to as Microbial Ecosystem Therapeutic-2 (MET-2).

In this open label, single center, multiple dose pilot study of 19 patients will be recruited. Patients will be given an initial daily loading dose of MET-2 over 2 days followed by a maintenance dose of MET-2 over 8 days. Patients experiencing treatment failure after the first dose may be offered a second, higher loading dose of MET-2. Patients failing the second loading dose of MET-2 may be offered a higher dose of MET-2 via colonoscopy.

The primary objective is clinical resolution of diarrhea with no CDI relapse at 30 days following the last dose of MET-2, i.e., absence of recurrence of diarrheal symptoms with laboratory-confirmed evidence of C. difficile 30 days after last dose of treatment.

The secondary objectives are: i) Safety and tolerability, including adverse events of grade 2 or above; ii) Overall well-being including number of bowel movements and energy level, etc. as based on standardized IBS questionnaire; iii) Presence of MET-2 bacteria in stool at 30 days, based on DNA sequencing; and, iv) Mortality, at end of follow up period - mortality attributable to CDI will also be determined, by performing a detailed clinical chart review on any patient who expires during the follow up period.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old.
2. Able to provide informed consent, or have a caregiver able to provide consent
3. Meets the definition of non-severe recurrent CDI (see Section 2.1, above) AND
4. Has had a positive stool test for C. difficile within 60 days of enrolment
5. Able to undergo colonoscopy and enemas
6. Not pregnant
7. Willing to participate in follow up as part of the study

In addition, the patient must agree to undergo stool testing and blood screening tests that are part of the study, including hepatitis and HIV testing

Exclusion Criteria:

1. Life expectancy < 6 months
2. Evidence of severe CDI ((neutropenia (ANC<1000) or WBC>30, creatinine >2X baseline, presence of toxic megacolon or intestinal perforation, admission to ICU)
3. History of chronic diarrhea
4. Need for regular use of agents that affect GI motility (narcotics such as codeine or morphine, agents such as loperamide or metoclopramide)
5. Use of antibiotics for another infection (other than CDI)
6. Colostomy
7. Elective surgery that will require preoperative antibiotics planned within 6 months of enrolment
8. Pregnant or planning to get pregnant in the next 6 months
9. Unable to tolerate MET-2 for any reason
10. Any condition for which colonoscopy or enema may be contraindicated (e.g., neutropenia, thrombocytopenia, bleeding disorders, severe colitis, etc)
11. Any condition for which, in the opinion of the investigator, the patient should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
To demonstrate clinical resolution of diarrhea with no CDI relapse, | 30 days
  To demonstrate clinical resolution of diarrhea with no CDI relapse at 30 days following the last dose of MET-2, the subject will undergo full physical examination including Blood Pressure, Heart rate and body temperature measurement. A blood test will be conducted with chemistry panel, and CBC with differential. Stool test and culture will also be conducted to measure the presence of C.difficile and DNA sequencing will determine the presence of MET-2 bacteria in the stool.

SECONDARY OUTCOMES:
Incidence of adverse events (safety and tolerability) | 3 months
  safety and tolerability, including adverse events of grade 2 or above
number of bowel movements (overall well-being) | 3 months
  overall well-being including number of bowel movements, etc as based on standardized IBS questionnaire
Presence of MET-2 bacteria | 30 days
  Presence of MET-2 bacteria in stool at 30 days, based on DNA sequencing
mortality | 3 months
  Mortality, at end of follow up period - mortality attributable to CDI will also be determined, by performing a detailed clinical chart review on any patient who expires during the follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Dina Kao, MD, Principal Investigator — University of Alberta, Edmonton Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kao D, Wong K, Franz R, Cochrane K, Sherriff K, Chui L, Lloyd C, Roach B, Bai AD, Petrof EO, Allen-Vercoe E. The effect of a microbial ecosystem therapeutic (MET-2) on recurrent Clostridioides difficile infection: a phase 1, open-label, single-group trial. Lancet Gastroenterol Hepatol. 2021 Apr;6(4):282-291. doi: 10.1016/S2468-1253(21)00007-8. Epub 2021 Feb 23. PMID 33631102